CLINICAL TRIAL: NCT04461509
Title: High-Resolution, 18F-PSMA PET-MRI for Mapping Prostate Cancer in Patients Considering Focal High-Intensity Focused Ultrasound (HIFU) Therapy or Radical Prostatectomy
Brief Title: High Resolution, 18F-PSMA PET-MRI Before Prostate Cancer HIFU or Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alessandro D'Agnolo (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Alessandro D'Agnolo, Co-Director Nuclear Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000832
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Disease
Keywords: Diagnostic imaging; High-Intensity Focused Ultrasound; HIFU; 18F-PSMA; high resolution diffusion-weighted imaging
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Neoplasms; Genital Diseases, Male; Prostatic Diseases | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Intervention Model Description: Patients are identified by investigator and enrolled in Arm 1 (HIFU) or Arm 2 (RP)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM 1 (HIFU) - 18F-PSMA (Experimental): 10 mCi ±20% F18-PSMA injection
  Interventions: Drug: 18F-PSMA
- ARM 2 (RP) - 18F-PSMA (Experimental): 10 mCi ±20% F18-PSMA injection
  Interventions: Drug: 18F-PSMA

INTERVENTIONS:
Drug: 18F-PSMA — Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-PSMA)
  Other Names:
  18F-DCFPyL Injection prostate-cancer-specific radiotracer
  Other Names: 18F-DCFPyL Injection

SUMMARY:
This prospective trial aims to determine if enhanced prostate imaging using two novel imaging technologies (high resolution DWI and 18F-PSMA PET-MRI) will detect prostate cancers not seen on standard multiparametric prostate MRI in patients considered candidates for focal HIFU.

DETAILED DESCRIPTION:
This is a prospective trial to evaluate the effectiveness of 18F-PSMA PET-hrMRI versus standard mpMRI at identifying prostate cancer targets for HIFU therapy.

Participants with clinically localized, unilateral high grade prostate cancer (Gleason score 7-10 prostate cancer localized to one lobe on prior biopsies) OR at high risk for having unrecognized high grade prostate cancer (overall Gleason score 6 with > half of systematic biopsy cores positive and > 50% of core involvement in at least one core), interested in HIFU would receive both a standard mpMRI and 18F-PSMA PET-hrMRI.

Participants would then undergo a mapping biopsy using a standard sextant template plus MRI/US-fusion targeted biopsy of any lesion suspicious lesion on mpMRI or PET-hrMRI.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy consisting of ≥ 10 tissue cores sampled
2. PSA <20 ng/mL (for HIFU arm only)
3. cT1-cT2c
4. Either overall Gleason score > 7 with Gleason grade 4 or 5 component localized to one lobe (i.e. right or left) OR overall Gleason score 6 with > half of systematic biopsy cores positive and > 50% of core involvement in at least one core (for HIFU arm only)
5. Patient considering focal HIFU therapy or robotic radical prostatectomy

Exclusion Criteria:

1. Previous local therapy for prostate cancer
2. Inability to receive PET tracer
3. Inability to receive MRI
4. Estimated glomerular filtration rate (GFR) <15 mL/min/1.73 m2
5. Any other condition which, in the investigator's option, may make the patient a poor candidate for participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D'Agnolo, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Basso Dias A, Ghai S, Ortega C, Mirshahvalad SA, Perlis N, Berlin A, Avery L, Veit-Haibach P, van der Kwast T, Metser U. Impact of 18F-DCFPyL PET/MRI in Selecting Men With Low-/Intermediate-Risk Prostate Cancer for Focal Ablative Therapies. Clin Nucl Med. 2023 Oct 1;48(10):e462-e467. doi: 10.1097/RLU.0000000000004819. PMID 37682613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial opened to accrual on 04/06/2021 with first subject enrolled on study 04/06/2021. Recruitment occurred at Cedars-Sinai Medical Center.
Groups:
- ARM 1 (HIFU) - 18F-PSMA; ARM 2 (RP) - 18F-PSMA: 10 mCi ±20% F18-PSMA injection
  18F-PSMA: Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-PSMA)
  Other Names:
  18F-DCFPyL Injection prostate-cancer-specific radiotracer
Period: Overall Study
Arm/Group | ARM 1 (HIFU) - 18F-PSMA | ARM 2 (RP) - 18F-PSMA
Started | 29 | 33
Completed | 24 | 32
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM 1 (HIFU) - 18F-PSMA | ARM 2 (RP) - 18F-PSMA | Total
Number analyzed (Participants) | 24 | 32 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 17 | 27
  >=65 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 32 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 22 | 28 | 50
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 15 | 23 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 32 | 56

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint (HIFU): Identification of New Cancers
Description: The grade of the cancer is assessed by biopsy prior to HIFU. Systematic and targeted prostate biopsies assess presence or absence of cancer in each zone of the prostate, including both systematic and targeted zones. Each zone with cancer is graded using the Gleason score (range 6-10, with higher scores associated with more aggressive disease). The primary outcome is for detection of any additional cancer with advanced imaging techniques of hrMRI or PSMA-PET MRI over standard multiparametric MRI. Any cancer is defined as "Gleason 6 or higher." We also did an exploratory analysis looking at detection of additional cancers with Gleason scores of 7 or higher.
Time Frame: At time of pre-HIFU biopsy
Population: The number of participants analyzed is 32 and not 29, because some participants switched over to the RP arm after already completing study intervention (imaging).
Measure: Number; unit: biopsy-proven cancerous zones
Units Other Than Participants: biopsy-zones
Groups:
- ARM 1 (HIFU) - 18F-PSMA: 10 mCi ±20% F18-PSMA injection
  18F-PSMA: Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-PSMA)
  Other Names:
  18F-DCFPyL Injection prostate-cancer-specific radiotracer
  Difference between sensitivities to identify prostate lesions.
Arm/Group | ARM 1 (HIFU) - 18F-PSMA
Number analyzed (Participants) | 32
Number analyzed (biopsy-zones) | 192
biopsy-proven cancerous zones
  Gleason 6+ | 85
  Gleason 7+ | 49

2. Primary Outcome: Primary Endpoint (Prostatectomy):
Description: To determine the sensitivity in detection of prostatic carcinoma of novel imaging modalities of hrMRI and/or F18-PSMA PET compared to reference standard mpMRI in patients scheduled to undergo radical prostatectomy.
Time Frame: preoperative PET-hrMRI prior to prostatectomy, less than 3 weeks before surgery
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Secondary Endpoint (HIFU):
Description: Negative biopsy rate on systematic and targeted biopsy 6 months following HIFU therapy. Data presented are from both systematic + targeted biopsy as a single unit. For example, a positive biopsy from a given area of the prostate could have come from either systematic or targeted cores.
Time Frame: 6 months following standard HIFU therapy
Population: Negative for any cancer in treated area, including high and low grade cancer 17/22 (77.3%) Negative for high-grade cancer in treated area 18/22 (81.8%)
  There were 4/22 patients who had high grade cancer in the treated area, and one patient who had low grade cancer in the treated area. Hence, 18/22 were negative for high grade cancer in the treated area while 17/22 were negative for both high grade or low grade cancer.
Measure: Count of Participants; unit: Participants
Groups:
- ARM 1 (HIFU) - 18F-PSMA: 10 mCi ±20% F18-PSMA injection
  18F-PSMA: Imaging (comparing standard and experimental high resolution diffusion-weighted imaging [DWI] MRI with 18F-PSMA)
  Other Names:
  18F-DCFPyL Injection prostate-cancer-specific radiotracer
  Negative biopsy rate on systematic and targeted biopsy 6 months following HIFU therapy.
Arm/Group | ARM 1 (HIFU) - 18F-PSMA
Number analyzed (Participants) | 22
Participants
  Negative for any cancer in treated area, including high and low grade cancer | 17
  Negative for high-grade cancer in treated area | 18

4. Secondary Outcome: Secondary Endpoint (Prostatectomy):
Description: Specificity of hrMRI, F18-PSMA PET and mpMRI for detecting all tumors and metastasis at 6 months follow up.
Time Frame: 6 months following standard HIFU therapy
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Exploratory Endpoint:
Description: RNAseq transcriptome analysis of lesions that are positive on mapping biopsy. Sensitivity and specificity of PET-hrMRI for detecting all tumors detected on prostatectomy pathology.
Time Frame: After study completion, an average of 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Arm/Group | ARM 1 (HIFU) - 18F-PSMA | ARM 2 (RP) - 18F-PSMA
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/24 | 4/32
Other Adverse Events (participants affected / at risk) | 3/24 | 5/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (HIFU) - 18F-PSMA (N=24) | ARM 2 (RP) - 18F-PSMA (N=32)
SOB (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sigmoid Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Wall Fluid Collection (Hepatobiliary disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Intractable Back Pain (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM 1 (HIFU) - 18F-PSMA (N=24) | ARM 2 (RP) - 18F-PSMA (N=32)
Acute DVT (Deep Vein Thrombosis) Right Femoral Vein (Vascular disorders) | 0 (0) | 1 (1)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Blood Loss Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Septecemia (Infections and infestations) | 0 (0) | 1 (1)
Syncope Post-Chemo (General disorders) | 0 (0) | 1 (1)
Fever Post-Chemo (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Abdominal Pain (General disorders) | 0 (0) | 1 (1)
Increased ALT (Alanine aminotransferase) (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Perineal Pain (General disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right Groin Pain (General disorders) | 1 (1) | 0 (0)
Hyponatremia (Nervous system disorders) | 1 (1) | 0 (0)
Bladder Discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)
Burning Urination for One Week (Renal and urinary disorders) | 1 (1) | 0 (0)
Facial Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis of Left Knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Effusion of Left Knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tongue Swelling - Allergic Reaction to Contrast (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04461509/Prot_SAP_000.pdf